CLINICAL TRIAL: NCT03199872
Title: A Phase I/II Study of RV001V, a RhoC Anticancer Vaccine, Against Metastasis From Solid Tumours
Brief Title: RV001V, a RhoC Anticancer Vaccine, Against Metastasis From Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RhoVac APS (Industry)
Collaborators: Dantrials Aps (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RhoVac-001
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: Prostatectomised cancer patients
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RV001V (Experimental): RV001 Vaccine 0.1 mg/mL (RV001V). RV001V consists of the peptide RV001 and the adjuvant Montanide ISA 51.
  Interventions: Biological: RV001V

INTERVENTIONS:
Biological: RV001V — Sc injection

SUMMARY:
The study will evaluate safety and immunological response to RhoC peptide vaccine in patients with prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients prostatectomised (PT) due to histologically verified adenocarcinoma of the prostate gland who currently are not being treated, or expected within the next 8 months to be treated, with any anti-cancer treatment.
* ECOG performance status 0 or 1.

Exclusion Criteria:

* Patient has been treated with Androgen Deprivation Therapy (ADT), or expected to receive such treatment within the next 8 months from enrolment.
* Severe medical conditions, such as but not limited to severe asthma/chronic obstructive pulmonary disease (COPD), New York Heart Association (NYHA) grading 3 or above, poorly regulated insulin dependent diabetes, any significant organ damage as judged by the Investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Sonne, MD, PhD, Principal Investigator — Dantrials Aps
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuhmacher J, Heidu S, Balchen T, Richardson JR, Schmeltz C, Sonne J, Schweiker J, Rammensee HG, Thor Straten P, Roder MA, Brasso K, Gouttefangeas C. Vaccination against RhoC induces long-lasting immune responses in patients with prostate cancer: results from a phase I/II clinical trial. J Immunother Cancer. 2020 Nov;8(2):e001157. doi: 10.1136/jitc-2020-001157. PMID 33184050

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: RV001V: RV001 Vaccine 0.1 mg/mL (RV001V). RV001V consists of the peptide RV001 and the adjuvant Montanide ISA 51.
  RV001V: A total of 11 s.c.injection with RV001V. The first 6 injections were given every 2 weeks, whereas the remaining 5 vaccinations were administered with 4 weeks between each injection.
Period: Overall Study
Arm/Group | Experimental: RV001V
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: RV001V: RV001 Vaccine 0.1 mg/mL (RV001V). RV001V consists of the peptide RV001 and the adjuvant Montanide ISA 51.
  RV001V: Sc injection
Arm/Group | Experimental: RV001V
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 22

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Participants With Treatment-related Adverse Events
Description: Proportions of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 8 month
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: RV001V
Number analyzed (Participants) | 22
Participants | 22

2. Secondary Outcome: Immunological Response
Description: RV001-specific immunological response after treatment from baseline to each treatment and follow-up
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: RV001V
Number analyzed (Participants) | 21
Participants | 18

ADVERSE EVENTS:
Time Frame: 20 months
Description: Non-TEAEs (Treatment Emergent Adverse Events) took place before the first vaccination.
  TEAEs took place after first vaccination and up to start of follow up phase (Visit 13). Only related AEs and SAEs are to be captured in the follow up period.
Arm/Group | Experimental: RV001V
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: RV001V (N=22)
Impaired healing (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: RV001V (N=22)
Injection site reaction (General disorders) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03199872/Prot_SAP_000.pdf